CLINICAL TRIAL: NCT04250701
Title: Investigation of Postural Control, Grip Strength and Body Posture in Children With Intellectual Disability and Dyslexia
Brief Title: Postural Control, Grip Strength and Body Posture in Children With Intellectual Disability and Dyslexia
Status: Completed | Type: Observational
Sponsor: Ahmet Emir (Other)
Responsible Party: Sponsor-Investigator, Ahmet Emir, Lecturer, Medipol University
Organization: Medipol University (Other)
Other Study IDs: 10840098-604.01.01-E.4231
Record Dates: First submitted 2020-01-28; First posted 2020-01-31 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Developmental Disability; Developmental Dyslexia; Intellectual Disability
Keywords: Postural Control,; Body Posture; Hand Grip
MeSH Terms: conditions — Developmental Disabilities; Dyslexia; Intellectual Disability

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Dyslexia (D)
  Interventions: Other: Body Posture Assessment
- Intellectual Disability (ID)
  Interventions: Other: Body Posture Assessment
- Control (C)
  Interventions: Other: Body Posture Assessment

INTERVENTIONS:
Other: Body Posture Assessment — Application of three evaluations above at a one time.
  Other Names: Postural Control Assessment; Hand Grip Strength Assessment

SUMMARY:
This study investigates physical changes in children with Dyslexia and Intellectual Disability. Participants divided into three groups and Body Posture, Postural Control and Hand Grip Strengths was evaluated.

DETAILED DESCRIPTION:
Children with Intellectual Disability and Dyslexia have academic and behavioral problems but also they might have physical changes related to poor motor development.

Three evaluation method was used in study. Postural Deformities were evaluated by PostureScreen Mobile App which is a mobile app allows to assess photographic body posture in four aspects (anterior, posterior, lateral) Postural Control was tested by Wii Balance Board. Wii balance board is a force plate that can measure person's center of gravity displacements Hand grip strength tested by Jamar Hand Dynamometer. It was completed according to American Hand Therapist's Association guidelines.

All data collected from participants have analysed within the control group (typical developed children)

ELIGIBILITY:
Inclusion Criteria:

1. no comorbid diagnosis alongside ID and Dyslexia (dysgraphia, dyscalculia, attention deficit hyperactivity disorder, etc.)
2. no orthopedic/physical disability

Exclusion Criteria

1. Presence of previous training for physical or motor development
2. Previous surgery.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Study population consisted children diagnosed with Dyslexia and Intellecutal Disability who continue their regular special education. The investigators also enrolled age matched typical developed children to establish control group
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2018-01-10 (Actual); Study Completion 2018-06-26 (Actual)

PRIMARY OUTCOMES:
Body Posture Assessment | through study completion, an average of 1 year
  It is a photographic body posture assessment done by mobile app. It shows deviations of certain body parts such as head, shoulder, pelvis towards to gravitational line.
Postural Control Evaluation | through study completion, an average of 1 year
  It is a wii balance board which can be used as a force plate. It tests displacements of Center of Pressure and Velocity of Center of Pressure and That gives an opinion about balance.
Hand Grip Strength | through study completion, an average of 1 year
  It is a basic force measurement of hand grip with dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Emir, Msc, Principal Investigator — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Beykoz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No